CLINICAL TRIAL: NCT02990390
Title: Shanghai First Maternity and Infant Hospital
Brief Title: The Epidemiology of Recurrent Spontaneous Abortion Associated With Thrombophilla
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Shihua Bao, Principal Investigator, Shanghai First Maternity and Infant Hospital
Other Study IDs: ShanghaiFMIH-0001
Record Dates: First submitted 2016-11-27; First posted 2016-12-13 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-11

CONDITIONS: Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
RSA is a multifactorial disorder resulting from genetic factors, anatomic factors, autoimmune disorders, endocrine dysfunction, thrombophilia, life style factors, and maternal infections. However, the underlying causes remain undetermined in up to 50% of cases. In this clinical cohort study, we intended to get an epidemiological evidence for patients with recurrent spontaneous abortion associated with thrombophilla.

ELIGIBILITY:
Inclusion Criteria:

* Woman who had 2 miscarriages before 12(th) week of gestation.Signed consent form.

Exclusion Criteria:

1. having experienced severe allergies, trauma history and/or operation history within 3 months;
2. with a history of mental illness and/or family history of mental illness
3. limb disabled
4. taking medicine within one month
5. suffering major events or having mood swings
6. with a history of recurrent pregnancy loss
7. having internal and surgical disease(after having variety of physical examination such as electrocardiogram/hepatic and renal function/blood routine and urine routine)
8. chromosome aberrations in anyone of the couple.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Woman who had their Second miscarriage before 12(th) week of gestation.
Sampling Method: Probability Sample
Enrollment: 45000 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
D-Dimer | through study completion, an average of 3 year

SECONDARY OUTCOMES:
BMI in kg/m^2 | through study completion, an average of 3 year
platelet aggregation time | through study completion, an average of 3 year
anticardiolipin antibody | through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided